CLINICAL TRIAL: NCT02530840
Title: Impact:Improving Adherence and Commitment to Treatment
Brief Title: Improving Adherence and Commitment to Treatment in Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clalit Health Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0025-14-COM
Record Dates: First submitted 2015-08-16; First posted 2015-08-21 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2016-07

CONDITIONS: Type 2 Diabetes
Keywords: imbalanced diabetic patients; HbA1c; peers
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- medical team (Experimental): personal meetings and follow-up of un-balanced diabetic patients by trained medical team (nurse and doctor), which designed to promote adherence to healthy life style and medical therapy.
  Interventions: Behavioral: medical team
- peers group (Experimental): group meetings and follow-up of un-balanced diabetic patients by trained peers (peers: balanced diabetic patients),which designed to promote adherence to healthy life style and medical therapy.
  Interventions: Behavioral: peers group
- SMS notifications (Experimental): un-balanced diabetic patients receiving daily SMS with content,which designed to promote adherence to healthy life style and medical therapy.
  Interventions: Behavioral: SMS notification
- control (No Intervention): un-balanced diabetic patients will get the basic and regular treatment for diabetic patients according to Clalit Health Services. In addition, the patients will have the same check-ups like all the patients in the experimental arms.

INTERVENTIONS:
Behavioral: medical team — Lowering HbA1c by behavioral changes in meetings with the medical team.
  Arms: medical team
Behavioral: peers group — Lowering HbA1c by behavioral changes in meetings with the peers group.
  Arms: peers group
Behavioral: SMS notification — Lowering HbA1c by behavioral changes in meetings with the SMS notification
  Arms: SMS notifications

SUMMARY:
In the IMPACT project, the investigators want to improve adherence and commitment to treatment.

DETAILED DESCRIPTION:
In this study the investigators use 3 interventions in diabetic patients and one control, to find what is the best intervention to improve adherence to healthy life style and medication therapy. the 3 intervention as followed: 1) meetings and follow-up by the medical team; 2) meetings and follow-up by trained peers; 3) system for sending SMS, operate according to algorithm.

ELIGIBILITY:
Inclusion Criteria:

1. type 2 diabetes
2. age 30-70
3. Oral medication or insulin
4. According to the HbA1c test result, 0.5% above the target for the patient's personal balance and below the 10%, the most recent, but in any event not more than six months prior to the study patient recruitment
5. BMI<35
6. Patients speak and read Hebrew
7. owners of a mobile phone that can receive text messages (SMS messages/ notifications) and have the ability to use the application (relevant for the SMS notification arm)

Exclusion Criteria:

1. Active malignant disease
2. creatinine levels above 2
3. Getting medicines that elevate sugar levels as steroids, chemotherapy
4. Three months after Myocardial Infraction (myocardial ischemia), surgical intervention, cardiac event
5. Patients who are planning major surgery
6. Patients who are planning a residential zone change
7. Patients with acute complications of diabetes under active treatment (such as limb amputation)
8. Patients diagnosed with unbalanced mental disorders
9. patients who can not sign the form on their own "informed consent"
10. patients suffering from dementia
11. Patients who are not mobile (dependent on the therapist)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-07 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Diabetes Control as Expressed by the Change in HbA1c % | 0, 6, 12 & 18 months
  Participants will undergo HbA1c periodical lab test, the data needed for the trial will be extracted from electronic medical record

CONTACTS AND LOCATIONS:
Overall Officials: Margalit Goldfracht, prof., Principal Investigator — Director of the Department of promoting quality of family medicine
Locations (1):
- Clalit Health Institute, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No